CLINICAL TRIAL: NCT04693078
Title: Detection of Colonic Polyps Via a Large Scale AI System
Brief Title: Detection of Colonic Polyps Via a Large Scale Artificial Intelligence (AI) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Google LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0309-19-SZMC
Record Dates: First submitted 2020-07-01; First posted 2021-01-05 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Colonic Polyp
Keywords: Colonoscopy Performance
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Consecutive patients undergoing screening or surveillance colonoscopy in whom a new polyp detection system based on deep learning will be used during the procedure.
  Interventions: Device: AI polyp detection system based on deep learning

INTERVENTIONS:
Device: AI polyp detection system based on deep learning — A Polyp detection system based on deep learning and artificial intelligence, which can alert the operator in real-time to the presence and location of polyps during a colonoscopy.

SUMMARY:
Colonoscopy is the gold standard for detection and removal of precancerous lesions, and has been amply shown to reduce mortality. However, the miss rate for polyps during colonoscopies is 22-28%, while 20-24% of the missed lesions are histologically confirmed precancerous adenomas. To address this shortcoming, the investigators propose a new polyp detection system based on deep learning, which can alert the operator in real-time to the presence and location of polyps during a colonoscopy. The investigators dub the system DEEP: (DEEP) DEtection of Elusive Polyps. The DEEP system was trained on 3,611 hours of colonoscopy videos derived from two sources, and was validated on a set comprising 1,393 hours of video, coming from a third, unrelated source. For the validation set, the ground truth labelling was provided by offline gastroenterologist annotators, who were able to watch the video in slow-motion and pause/rewind as required; two or three specialist annotators examined each video.

This is a prospective, non-blinded, non-randomized pilot study of patients undergoing elective screening and surveillance colonoscopies using DEEP.

The aim of the study is to:

Assess the:

1. Number of additional polyps detected by the DEEP system in real time colonoscopy.
2. Safety by prospective assessment of the rate of adverse events during the study period attributed or not to the use of the DEEP system.
3. Stability of the DEEP system by measuring the rate of false positives (False Alarms) per colonoscopies 4 And to examine its feasibility and usefulness of in clinical practice by assessing the colonoscopist user experience while using the DEEP system in a 5 point scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects undergoing routine screening or surveillance colonoscopy in an ambulatory non urgent setting.
* Able to understand the study protocol and sign inform consent.

Exclusion Criteria:

* Previous surgery involving the colon or rectum
* Known diagnosis of colorectal cancer
* Known history of inflammatory bowel disease
* Known or suspected diagnosis of familial polyposis syndrome

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Diseases Institute, Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be shared only on request and after consent form the patient and the institutional ethics committee

REFERENCES:
- [Derived] Livovsky DM, Veikherman D, Golany T, Aides A, Dashinsky V, Rabani N, Ben Shimol D, Blau Y, Katzir L, Shimshoni I, Liu Y, Segol O, Goldin E, Corrado G, Lachter J, Matias Y, Rivlin E, Freedman D. Detection of elusive polyps using a large-scale artificial intelligence system (with videos). Gastrointest Endosc. 2021 Dec;94(6):1099-1109.e10. doi: 10.1016/j.gie.2021.06.021. Epub 2021 Jun 30. PMID 34216598

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Israel | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Additional Polyps Detected by the DEEP System in Real Time Colonoscopy
Description: During the colonoscopy procedure, in real time when a polyp is found, the colonoscopist will rate the polyp as an elusive polyp detected by the system that might have been missed or a polyp that would have been detected with or without the system.
  The outcome measure will be reported as the average of additional polyps detected per colonoscopy by the DEEP system
Time Frame: Through study completion, an average of 12 months
Measure: Mean (95% Confidence Interval); unit: Added polyps detected per colonoscopy
Arm/Group | Intervention Arm
Number analyzed (Participants) | 100
Added polyps detected per colonoscopy | 0.89 [0.66 to 1.12]

2. Primary Outcome: The Rate of Adverse Events During the Study Attributed or Not to the Use of the DEEP System
Description: Prospective assessment adverse events during the study. The following adverse event will be monitored: Perforation, bleeding, and cardiorespiratory adverse events during the procedure
Time Frame: Until discharge, assessed up to 7 days
Measure: Number; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 100
Participants | 0

3. Secondary Outcome: Rate of False Positives (False Alarms) Per Colonoscopy
Description: During the colonoscopy procedure, in real time after each polyp found by the DEEP system, the colonoscopist will rate the polyp as either a true polyp or a false positive detection or a "false alarm" this measure will be reported as the average of false positive detection per colonoscopy
Time Frame: Through study completion, an average of 12 months
Measure: Mean (95% Confidence Interval); unit: False positive alarms per colonoscopy
Arm/Group | Intervention Arm
Number analyzed (Participants) | 100
False positive alarms per colonoscopy | 3.87 [3.34 to 4.40]

4. Secondary Outcome: Colonoscopist User Experience While Using the DEEP System in a 5 Point Scale
Description: At the end of the procedures the colonoscopist will be requires to answer the question "from a scale of 1-5 how useful did you find the system in this procedure?", where higher scores represent more usefulness. This measure will be reported as the average score form all 100 procedures.
Time Frame: Through study completion, an average of 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 100
score on a scale | 3.9 [3.7 to 4.1]

ADVERSE EVENTS:
Time Frame: 6 months after the end of the study
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT04693078/Prot_SAP_000.pdf